CLINICAL TRIAL: NCT00555880
Title: A Multi-Center, Double-Blind, Randomized, Placebo-controlled, Crossover Study to Assess the Clinical Benefit of Midodrine Hydrochloride in Subjects With Moderate to Severe Neurogenic Orthostatic Hypotension
Brief Title: Study to Assess the Benefit of Midodrine in the Treatment of Patients With Neurogenic Orthostatic Hypotension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD426-404
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Hypotension, Orthostatic
MeSH Terms: conditions — Hypotension, Orthostatic | interventions — Midodrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Midodrine hydrochloride
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Midodrine hydrochloride — one dose, 10-30mg, given orally
  Other Names: ProAmatine
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
The purpose of this clinical study is to evaluate the clinical effect of midodrine hydrochloride (ProAmatine®) compared to placebo in patients with orthostatic hypotension by measuring the time to onset of near syncopal symptoms and assessing several cardiovascular measurements, such as heart rate, blood pressure, and ECG, using the tilt table test.

ELIGIBILITY:
Inclusion Criteria:

* The male or female subjects must be 18 years of age or older and ambulatory. (Subjects must not require assistance with a walker or wheelchair to perform regular daily activities at all times.)
* Women of childbearing potential must have a negative serum beta HCG pregnancy test at screening and baseline.
* The subject has been diagnosed with symptomatic orthostatic hypotension due to Parkinson's disease, multiple system atrophy, pure autonomic failure or autonomic neuropathy (i.e. neurogenic orthostatic hypotension).
* The subject manifests one of the following symptoms while standing or has a history of one of the following when not treated for orthostatic hypotension: dizziness, lightheadedness, feeling faint or feeling like they may black out.
* The subject is willing and able to undergo the procedures required by this protocol including morning office visits, assessment completion, protocol compliance and participation in the wash-out period.
* The subject has signed an Institutional-Review-Board approved written informed consent form prior to any study procedures taking place.

Exclusion Criteria:

* The subject is a pregnant or lactating female.
* The subject has pre-existing sustained supine hypertension greater than 180 mm Hg systolic and 110 mm Hg diastolic.
* The subject is taking medications such as vasodilators, pressors, diuretics, ACE inhibitors, angiotensin receptor blockers, beta-blockers, combined alpha and beta-blockers, MAOI's, herbals or specific mixed effect medications.
* The Principal Investigator deems any laboratory test abnormality clinical significant.
* The subject has a diagnosis of any of the following disorders at the time of screening: pheochromocytoma; cardiac conditions including: congestive heart failure within the previous 6 months, myocardial infarction within the previous 6 months, symptomatic coronary artery disease, history of ventricular tachycardia, or uncontrolled cardiac arrhythmias; thyrotoxicosis; uncontrolled diabetes mellitus (uncontrolled defined as a HgbA1c greater than or equal to 10%); history of cerebrovascular accident, transient ischemic attack (TIA) or symptomatic carotid artery stenosis within the previous 6 months; history of coagulopathies; pulmonary hypertension; severe psychiatric disorders; renal failure (Creatinine equal to or greater than 2 times the upper limit of normal)
* The subject has a concurrent chronic or acute illness, disability, or other condition that might confound the results of the tests and/or measurements administered in this trial, or that might increase the risk to the subject.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-09-08 (Actual); Primary Completion 2005-03-21 (Actual); Study Completion 2005-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (11):
- United States (11):
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Minnesota VA Medical Center, Minneapolis, Minnesota
  - Forest Park Neurophysiology, St Louis, Missouri
  - Mount Sinai Medical Center, New York, New York
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Absher Neurology, PA, Greenville, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Diabetes and Glandular Disease research Associates, PA, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Midodrine/Placebo: Participants received a single oral dose of Midodrine hydrochloride (HCl) followed by matching Placebo the next day
- Placebo/Midodrine: Participants received Placebo followed by a single oral dose of Midodrine HCl the next day
Period: Treatment Period 1 (1 Day)
Arm/Group | Midodrine/Placebo | Placebo/Midodrine
Started | 13 | 11
Completed | 13 | 11
Not Completed | 0 | 0
Period: Washout (1 Day)
Arm/Group | Midodrine/Placebo | Placebo/Midodrine
Started | 13 | 11
Completed | 13 | 11
Not Completed | 0 | 0
Period: Treatment Period 2 (1 Day)
Arm/Group | Midodrine/Placebo | Placebo/Midodrine
Started | 13 | 11
Completed | 13 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety and Full Analysis Set (FAS) populations, defined as all participants who received at least one dose of investigational product (Safety) and all participants who were randomized, received at least one dose of investigational product, and had at least one measurement of the time to near syncope during a tilt table test (FAS).
Groups:
- Midodrine/Placebo: Participants received a single oral dose of Midodrine HCl followed by matching Placebo the next day
- Placebo/Midodrine: Participants received matching Placebo followed by a single oral dose of Midodrine HCl the next day
- Total: Total of all reporting groups
Arm/Group | Midodrine/Placebo | Placebo/Midodrine | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (17.84) | 60.8 (12.91) | 60.0 (15.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 11 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 11 | 10 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Onset of Near-syncopal Symptoms During Tilt Table Testing
Description: The tilt table test is a 10-minute assessment performed using a manual or automated tilt table in a specialized laboratory. Subjects were moved onto the horizontal table and secured to the table with straps to prevent injury. After an equilibration period of at least 10 minutes with the subject at rest, the test began and the head of the tilt table was elevated to a 70-degree angle over a period of up to 30 seconds. The head-up tilt table test in this study was conducted 1 hour after administration of the study medication. The endpoint was a confirmed report of a near-syncopal symptom(s) (of sufficient severity that caused the patient to ask that the tilt table be returned to the horizontal position). Symptoms of near syncope were defined as dizziness, lightheadedness, feeling faint, or feeling like the subject might black out.
Time Frame: 1 hour post-dose
Population: The Full Analysis Set (FAS), defined as subjects who were randomized, received at least one dose of study drug, and had at least one measurement of time to syncope during tilt table testing.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Midodrine HCl: Midodrine HCl: one dose, 10-30mg, given orally
- Placebo: Placebo: A daily dose of Placebo tablets matching Midodrine HCl in appearance and number
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 24 | 24
seconds | 551.3 (115.63) | 461.0 (190.74)
Statistical Analysis 1: Comparison: Midodrine HCl vs Placebo; Test type: Superiority or Other; p = 0.1460, Sign test; Sign Statistic = 3.0 — Sign test was performed per analysis plan

2. Secondary Outcome: Time to Onset of Near-syncopal Symptoms in The Per-protocol Population
Description: as for outcome 1
Time Frame: 1 hour post-dose
Population: The Per-protocol set, defined as participants in the Full Analysis Set who completed the study and were protocol compliant.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 21 | 21
seconds | 544.3 (122.34) | 447.9 (199.31)
Statistical Analysis 1: Comparison: Midodrine HCl vs Placebo; Test type: Superiority or Other; p = 0.2266, Sign test; Sign statistic = 2.5 — Sign test was performed per analysis plan

3. Secondary Outcome: Time to Onset of Near-syncopal Symptoms in The Per-protocol Population Analysis #2
Description: The tilt table test is a 10-minute assessment performed using a manual or automated tilt table in a specialized laboratory. Subjects were moved onto the horizontal table and secured to the table with straps to prevent injury. After an equilibration period of at least 10 minutes with the subject at rest, the test began and the head of the tilt table was elevated to a 70-degree angle over a period of up to 30 seconds. The head-up tilt table test in this study was conducted 1 hour after administration of the study medication. The endpoint was a confirmed report of a near- syncopal symptom(s) (of sufficient severity that caused the patient to ask that the tilt table be returned to the horizontal position). Symptoms of near syncope were defined as dizziness, lightheadedness, feeling faint, or feeling like the subject might black out. In this outcome measure, the data analyzed are the same as for Outcome Measure 4 but the summary data are presented as least squares mean (standard error).
Time Frame: 1 hour post-dose
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 21 | 21
seconds | 545.1 (36.90) | 447.2 (36.90)
Statistical Analysis 1: Comparison: Midodrine HCl vs Placebo; Analysis of treatment difference; Test type: Superiority or Other; p = 0.0418, ANOVA — The P-value is based on type III sum of squares for treatment group from a mixed effect ANOVA model with sequence, period and treatment as fixed effects, and subject within sequence as a random effect; Least squares mean = 97.9 — Least squares mean for treatment difference (Midodrine HCL-Placebo)

4. Secondary Outcome: Time to Near-syncopal Symptoms at Treatment Visit 1
Description: as for outcome 1
Time Frame: 1 hour post-dose
Population: The Full Analysis Set, defined as subjects who were randomized, received at least one dose of study drug, and had at least one measurement of time to syncope during tilt table testing.
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 13 | 11
seconds | 539.5 (45.91) | 448.4 (49.91)
Statistical Analysis 1: Comparison: Midodrine HCl vs Placebo; Test type: Superiority or Other; p = 0.1928, ANOVA — The P-value is based on type III sum of squares for treatment group from a one-way ANOVA model; Least squares mean = 91.1 — Least squares mean for treatment difference (Midodrine HCL-Placebo)

5. Secondary Outcome: Duration of The Effect of Treatment at 3 Hours Post-dose
Description: Duration of effect was defined as the difference in time to onset of near-syncopal symptoms between the first and second tilt table test, conducted at 1 hour and 3 hours post-dose, respectively, at Treatment Visit 2 (time to onset at 3 hours minus time at 1 hour). The tilt table test is a 10-minute assessment performed using a manual or automated tilt table in a specialized laboratory. Subjects were moved onto the horizontal table and secured to the table with straps to prevent injury. After an equilibration period of at least 10 minutes with the subject at rest, the test began and the head of the tilt table was elevated to a 70-degree angle over a period of up to 30 seconds. The endpoint was a confirmed report of a near-syncopal symptom(s) (of sufficient severity that caused the patient to ask that the tilt table be returned to the horizontal position). Symptoms of near syncope were defined as dizziness, lightheadedness, feeling faint, or feeling like the subject might black out.
Time Frame: 1 and 3 hours post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 11 | 13
seconds | 45.1 (94.03) | 48.0 (114.96)
Statistical Analysis 1: Comparison: Midodrine HCl vs Placebo; Test type: Superiority or Other; p = 0.9479, t-test, 2 sided — The P-value is from a 2-sample t-test for difference in mean

6. Secondary Outcome: Total Score of the Orthostatic Hypotension Symptom Assessment (OHSA)
Description: The OHSA measures the severity of six symptoms/symptom complexes associated with orthostatic hypotension. Subjects rated symptoms experienced during the tilt table test on an eleven-point scale from "none" to "worst possible". The OHSA total score is the sum of six subscales, ranging from 0 (no symptoms) to 60 (worst possible symptoms). The OHSA was completed after the tilt table test was over, but was answered with reference to symptoms experienced during testing. The tilt table test is a 10-minute assessment performed using a manual or automated tilt table in a specialized laboratory. Subjects were moved onto the horizontal table and secured to the table with straps to prevent injury. After an equilibration period with the subject at rest, the test began and the head of the tilt table was elevated to a 70-degree angle over a period of up to 30 seconds. Symptoms of near syncope were defined as dizziness, lightheadedness, feeling faint, or feeling like the subject might black out.
Time Frame: Approximately 1 hour post-dose
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 24 | 24
scores on a scale | 13.7 (2.95) | 19.4 (2.95)
Statistical Analysis 1: Comparison: Midodrine HCl vs Placebo; Analysis of treatment; Test type: Superiority or Other; p = 0.0590, ANOVA — The P-value is based on type III sum of squares for treatment group from a mixed effect ANOVA model with sequence, period, and treatment as fixed effects and subject within sequence as a random effect; Least squares mean = -5.7 — Least squares mean for treatment difference (Midodrine HCl - Placebo)

7. Secondary Outcome: Scores for 6 Items of The OHSA
Description: The OHSA measures the severity of six symptoms/symptom complexes associated with OH: dizziness, lightheadedness, and feeling faint; problems with vision; weakness; fatigue; trouble concentrating; and head/neck discomfort. Subjects rated symptoms experienced during the tilt table test on an eleven-point scale from "none" to "worst possible". Scores for each subscale range from 0 (no symptoms) to 10 (worst possible symptoms). The OHSA was completed after the tilt table test was over, but was answered with reference to symptoms experienced during testing. The tilt table test is a 10-minute assessment performed using a tilt table in a specialized laboratory. Subjects were moved onto the horizontal table and secured with straps to prevent injury. After an equilibration period with the subject at rest, the test began and the head of the tilt table was elevated to a 70-degree angle over 30 seconds. Symptoms of near syncope were defined as dizziness, lightheadedness, and feeling faint.
Time Frame: Approximately 1 hour post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 24 | 24
scores on a scale
  Dizziness, Lightheadedness, and Feeling Faint | 3.4 (3.44) | 4.7 (3.57)
  Problems with Vision | 1.5 (2.32) | 2.7 (3.43)
  Weakness | 3.0 (3.13) | 4.1 (3.17)
  Fatigue | 2.7 (3.22) | 3.5 (3.48)
  Trouble Concentrating | 1.7 (2.04) | 2.6 (3.13)
  Head/Neck Discomfort | 1.9 (2.52) | 2.1 (3.21)
Statistical Analysis 1: Comparison: Midodrine HCl vs Placebo; Item Dizziness, Lightheadedness, and Feeling Faint-Analysis of treatment; Test type: Superiority or Other; p = 0.0633, ANOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Midodrine HCl vs Placebo; Item Problems with Vision-Analysis of treatment; Test type: Superiority or Other; p = 0.0191, ANOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Midodrine HCl vs Placebo; Item Weakness-Analysis of treatment; Test type: Superiority or Other; p = 0.0727, ANOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Midodrine HCl vs Placebo; Item Fatigue-Analysis of treatment; Test type: Superiority or Other; p = 0.2820, ANOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Midodrine HCl vs Placebo; Item Trouble Concentrating-Analysis of treatment; Test type: Superiority or Other; p = 0.0880, ANOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Midodrine HCl vs Placebo; Item Head/Neck Discomfort-Analysis of treatment; Test type: Superiority or Other; p = 0.6439, ANOVA — [p-value comment as in outcome 6, analysis 1]

8. Secondary Outcome: Number of Participants With Improvement of Clinician Clinician's Global Impression- Improvement (CGI-I) Scores After Tilt Table Test
Description: The CGI-I instrument assesses the overall impression of the subject's orthostatic hypotension during the tilt table test by using a 7-point scale, with 1 being Very much improved; 2, Much improved; 3, Slightly improved; 4, No change; 5, Slightly worse; 6, Much worse; and 7, Very much worse. The clinician completed the CGI-I after each of the tilt table tests. A patient was assessed as "Improved" if the score was 1, 2, or 3. The tilt table test is a 10-minute assessment performed using a manual or automated tilt table in a specialized laboratory. Subjects were moved onto the horizontal table and secured to the table with straps to prevent injury. After an equilibration period of at least 10 minutes with the subject at rest, the test began and the head of the tilt table was elevated to a 70-degree angle over a period of up to 30 seconds. Symptoms of near syncope were defined as dizziness, lightheadedness, feeling faint, or feeling like the subject might black out.
Time Frame: 1 and 3 hours post-dose
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 24 | 24
participants
  Treatment Visit 1- 1 hour post-dose, n=13, 11 | 4 | 4
  Treatment Visit 2- 1 hour post-dose, n=11, 13 | 6 | 4
  Treatment Visit 2- 3 hour post-dose, n= 11, 12 | 3 | 5

9. Secondary Outcome: Number of Participants With Improvement of Patient CGI-I Scores After Tilt Table Test
Description: The CGI-I instrument assesses the overall impression of the subject's orthostatic hypotension during the tilt table test by using a 7-point scale, with 1 being Very much improved; 2, Much improved; 3, Slightly improved; 4, No change; 5, Slightly worse; 6, Much worse; and 7, Very much worse. The patient completed the CGI-I after each of the tilt table tests. A patient was assessed as "Improved" if the score was 1, 2, or 3. The tilt table test is a 10-minute assessment performed using a manual or automated tilt table in a specialized laboratory. Subjects were moved onto the horizontal table and secured to the table with straps to prevent injury. After an equilibration period of at least 10 minutes with the subject at rest, the test began and the head of the tilt table was elevated to a 70-degree angle over a period of up to 30 seconds. Symptoms of near syncope were defined as dizziness, lightheadedness, feeling faint, or feeling like the subject might black out.
Time Frame: 1 and 3 hours post-dose
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 24 | 24
participants
  Treatment Visit 1-1 hour post-dose, n= 13, 11 | 3 | 2
  Treatment Visit 2-1 hour post-dose, n= 11, 13 | 5 | 3
  Treatment Visit 2-3 hour post-dose, n= 11, 12 | 3 | 3

10. Secondary Outcome: Final Blood Pressure During Tilt Table Testing
Description: Blood pressure was recorded just before tilt table testing and immediately after. Timed readings were stopped once a subject experienced near-syncopal symptoms, except for subjects for whom the table was returned to horizontal before 1 minute; for these subjects, a reading was made at 1 minute and was included in analyses. The tilt table test is a 10-minute assessment performed using a manual or automated tilt table in a specialized laboratory. Subjects were moved onto the horizontal table and secured to the table with straps to prevent injury. After an equilibration period of at least 10 minutes with the subject at rest, the test began and the head of the tilt table was elevated to a 70-degree angle over a period of up to 30 seconds. Symptoms of near syncope were defined as dizziness, lightheadedness, feeling faint, or feeling like the subject might black out.
Time Frame: 1 hour post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 24 | 24
mmHg
  Systolic Pressure | 106.5 (37.27) | 90.2 (24.17)
  Diastolic Pressure | 70.6 (16.44) | 60.6 (15.04)
Statistical Analysis 1: Comparison: Midodrine HCl vs Placebo; Final systolic pressure-Analysis of treatment; Test type: Superiority or Other; p = 0.0378, ANOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Midodrine HCl vs Placebo; Final diastolic pressure-Analysis of treatment; Test type: Superiority or Other; p = 0.0108, ANOVA

11. Secondary Outcome: Systolic Blood Pressure at 1 Minute and 10 Minutes Into The Tilt Table Test Conducted 1 and 3 Hours Post-dose at Treatment Visit 2
Description: Blood pressure was recorded just before tilt table testing, at each minute during tilt table testing, and immediately after. Timed readings were stopped once a subject experienced near-syncopal symptoms, except for subjects for whom the table was returned to horizontal before 1 minute; for these subjects, a reading was made at 1 minute and was included in analyses. The tilt table test is a 10-minute assessment performed using a manual or automated tilt table in a specialized laboratory. Subjects were moved onto the horizontal table and secured to the table with straps to prevent injury. After an equilibration period of at least 10 minutes with the subject at rest, the test began and the head of the tilt table was elevated to a 70-degree angle over a period of up to 30 seconds. Symptoms of near syncope were defined as dizziness, lightheadedness, feeling faint, or feeling like the subject might black out.
Time Frame: 1 and 3 hours post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 24 | 24
mmHg
  At 1 minute 1 hour post-dose, n= 11, 13 | 142.2 (44.20) | 97.3 (24.55)
  At 1 minute 3 hours post-dose, n= 11, 12 | 110.1 (19.06) | 94.9 (31.36)
  At 10 minutes 1 hour post-dose, n= 10, 8 | 121.7 (37.57) | 102.9 (21.03)
  At 10 minutes 3 hours post-dose, n= 7, 6 | 108.3 (30.48) | 107.2 (19.32)

12. Primary Outcome: Time to Onset of Near-syncopal Symptoms During Tilt Table Testing Analysis #2
Description: The tilt table test is a 10-minute assessment performed using a manual or automated tilt table in a specialized laboratory. Subjects were moved onto the horizontal table and secured to the table with straps to prevent injury. After an equilibration period of at least 10 minutes with the subject at rest, the test began and the head of the tilt table was elevated to a 70-degree angle over a period of up to 30 seconds. The head-up tilt table test in this study was conducted 1 hour after administration of the study medication. The endpoint was a confirmed report of a near- syncopal symptom(s) (of sufficient severity that caused the patient to ask that the tilt table be returned to the horizontal position). Symptoms of near syncope were defined as dizziness, lightheadedness, feeling faint, or feeling like the subject might black out. In this outcome measure, the data analyzed are the same as for Outcome Measure 1 but the summary data are presented as least squares mean (standard error).
Time Frame: 1 hour post-dose
Population: The FAS, defined as subjects who were randomized, received at least one dose of study drug, and had at least one measurement of time to syncope during tilt table testing.
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 24 | 24
seconds | 552.4 (32.93) | 460.0 (32.93)
Statistical Analysis 1: Comparison: Midodrine HCl vs Placebo; Analysis of treatment difference; Test type: Superiority or Other; p = 0.0296, ANOVA — [p-value comment as in outcome 6, analysis 1]; Least squares mean = 92.4 — Least squares mean for treatment difference (Midodrine HCl - Placebo)

13. Secondary Outcome: Diastolic Blood Pressure at 1 Minute and 10 Minutes Into The Tilt Table Test Conducted 1 and 3 Hours Post-dose at Treatment Visit 2
Description: as for outcome 11
Time Frame: 1 and 3 hours post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 24 | 24
mmHg
  At 1 minute 1 hour post-dose, n= 11, 12 | 81.5 (19.09) | 60.8 (13.99)
  At 10 minutes 1 hour post-dose, n= 10, 8 | 79.6 (16.18) | 64.9 (11.22)
  At 1 minute 3 hours post-dose, n= 11, 12 | 66.1 (9.66) | 60.3 (18.53)
  At 10 minutes 3 hours post-dose, n= 7, 6 | 69.3 (13.55) | 60.7 (14.69)

14. Secondary Outcome: Heart Rate at 1 Minute and 10 Minutes Into The Tilt Table Test Conducted 1 and 3 Hours Post-dose at Treatment Visit 2
Description: Heart rate was recorded just before tilt table testing, at each minute during tilt table testing, and immediately after. Timed readings were stopped once a subject experienced near-syncopal symptoms, except for subjects for whom the table was returned to horizontal before 1 minute; for these subjects, a reading was made at 1 minute and was included in analyses. The tilt table test is a 10-minute assessment performed using a manual or automated tilt table in a specialized laboratory. Subjects were moved onto the horizontal table and secured to the table with straps to prevent injury. After an equilibration period of at least 10 minutes with the subject at rest, the test began and the head of the tilt table was elevated to a 70-degree angle over a period of up to 30 seconds. Symptoms of near syncope were defined as dizziness, lightheadedness, feeling faint, or feeling like the subject might black out.
Time Frame: 1 and 3 hours post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 24 | 24
beats per minute
  At 1 minute 1 hour post-dose, n= 11, 13 | 77.6 (13.93) | 80.5 (14.07)
  At 10 minutes 1 hour post-dose, n= 10, 8 | 77.7 (16.08) | 79.5 (16.48)
  At 1 minute 3 hours post-dose, n= 11, 12 | 79.7 (11.30) | 80.9 (13.19)
  At 10 minutes 3 hours post-dose, n= 8, 6 | 80.9 (11.66) | 81.3 (20.16)

15. Secondary Outcome: Number of Participants With Shifts in Reference to Normal Range For Hematology Analytes at Discharge
Description: For hematology, blood samples (5.0mL) were taken at screening, study admission (if greater than 14 days since screening) and discharge/early termination. The following parameters were assessed: hemoglobin, hematocrit, red blood cells (RBC), mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), white blood cell count - total and differential (WBC), and platelet count. A shift in reference to normal was either lower or higher at discharge.
Time Frame: Baseline to discharge
Population: The Safety population, defined as all subjects who received at least one dose of investigational product.
Measure: Number; unit: participants
Groups:
- All Participants: All randomized participants
Arm/Group | All Participants
Number analyzed (Participants) | 24
participants
  Hemoglobin | 1
  Hematocrit | 0
  RBC | 0
  MCV | 0
  MCH | 0
  MCHC | 2
  WBC | 1
  Platelet count | 0

16. Secondary Outcome: Number of Participants With Shifts in Reference to Normal Range For Clinical Chemistry at Discharge
Description: For biochemistry, blood samples (10.0mL) were taken at screening, admission (if greater than 14 days since screening) and discharge/early termination. The following parameters were assessed: sodium, potassium, calcium, blood urea nitrogen (BUN)/Urea, creatinine, albumin, total protein and albumin/globulin (A/G) ratio, globulin, aspartate transaminase (AST), alanine transaminase (ALT), alkaline phosphatase (ALP), gamma glutamyl transferase (GGT), total bilirubin, glucose, chloride, and creatine kinase. A shift in reference to normal was either lower or higher at discharge.
Time Frame: Baseline to discharge
Population: The Safety population, defined as all subjects who received at least one dose of investigational product.
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 24
participants
  Sodium | 0
  Potassium | 2
  Calcium | 1
  BUN/Urea | 0
  Creatinine | 1
  Albumin | 0
  Total protein and A/G ratio | 2
  Globulin | 0
  ALT | 0
  AST | 0
  ALP | 1
  GGT | 0
  Total bilirubin | 1
  Glucose | 6
  Chloride | 0
  Creatine kinase | 1

17. Primary Outcome: Time to Onset of Near-syncopal Symptoms During Tilt Table Testing-Re-analysis With The Koch Procedure
Description: The tilt table test is a 10-minute assessment performed using a manual or automated tilt table in a specialized laboratory. Subjects were moved onto the horizontal table and secured to the table with straps to prevent injury. After an equilibration period of at least 10 minutes with the subject at rest, the test began and the head of the tilt table was elevated to a 70-degree angle over a period of up to 30 seconds. The head-up tilt table test in this study was conducted 1 hour after administration of the study medication. The endpoint was a confirmed report of a near-syncopal symptom(s) (of sufficient severity that caused the patient to ask that the tilt table be returned to the horizontal position). Symptoms of near syncope were defined as dizziness, lightheadedness, feeling faint, or feeling like the subject might black out. The Koch procedure is a 3-step process to analyze results while utilizing the available information on magnitude of differences.
Time Frame: 1 hour post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Midodrine HCl | Placebo
Number analyzed (Participants) | 24 | 24
seconds | 551.3 (115.63) | 461.0 (190.74)
Statistical Analysis 1: Comparison: Midodrine HCl vs Placebo; Analysis of treatment; Test type: Superiority or Other; p = 0.0342, Signed Rank Test

18. Secondary Outcome: Number of Participants With Shifts in Reference to Normal Range For Urinalysis at Discharge
Description: For urinalysis, samples were taken at screening, study admission (if greater than 14 days since screening) and discharge/early termination): glucose, blood, protein, pH, specific gravity, leukocyte esterase, and microscopic examination. A shift in reference to normal was higher at discharge.
Time Frame: Baseline to discharge
Population: The Safety population, defined as all subjects who received at least one dose of investigational product.
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 24
participants
  Glucose | 1
  Blood | 2
  Protein | 0
  pH | 0
  Specific gravity | 0
  Leukocyte esterase | 2
  Microscopic examination | 0

ADVERSE EVENTS:
Description: Adverse events are reported by randomized arm and not by actual treatment intervention received.
Groups:
- Midodrine/Placebo: Participants received a single oral dose of Midodrine HCl (10-30mg) followed by placebo the next day.
- Placebo/Midodrine: Participants received Placebo followed by a single oral dose of Midodrine HCl (10-30mg) the next day.
Arm/Group | Midodrine/Placebo | Placebo/Midodrine
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/11
Other Adverse Events (participants affected / at risk) | 3/13 | 2/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Midodrine/Placebo (N=13) | Placebo/Midodrine (N=11)
Multiple sclerosis aggravated (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Midodrine/Placebo (N=13) | Placebo/Midodrine (N=11)
Nausea (Gastrointestinal disorders) | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Vomiting NOS (Gastrointestinal disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache NOS (Nervous system disorders) | 1 | 0
Hypertension aggravated (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.